CLINICAL TRIAL: NCT06818526
Title: A Randomized, Double-Blind, Placebo-Controlled, Two-Period Crossover Study to Evaluate the Efficacy and Safety of Huandao Conditioning Application in Adults with Allergic Rhinitis
Brief Title: Huandao Conditioning Application for Allergic Rhinitis Treatment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB113-209-A
Record Dates: First submitted 2025-02-05; First posted 2025-02-10 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Allergic Rhinitis
Keywords: allergic rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo Huandao Conditioning Application (Placebo Comparator)
  Interventions: Device: Placebo Huandao Conditioning App
- Therapeutic Huandao Conditioning Application (Experimental)
  Interventions: Device: Huandao Conditioning Application

INTERVENTIONS:
Device: Huandao Conditioning Application — Mobile Application Intervention: Huandao Conditioning App for Allergic Rhinitis Treatment
  Type: Software Application (Mobile App) Purpose: Energy balancing therapy based on traditional Chinese medicine meridian theory Application Method: Self-administered via smartphone Duration: 5-10 minutes per session
  Arms: Therapeutic Huandao Conditioning Application
Device: Placebo Huandao Conditioning App — Mobile Application Intervention: Placebo Huandao Conditioning App for Allergic Rhinitis Treatment
  Type: Software Application (Mobile App) Purpose: Energy balancing therapy based on traditional Chinese medicine meridian theory Application Method: Self-administered via smartphone Duration: 5-10 minutes per session
  Arms: Placebo Huandao Conditioning Application

SUMMARY:
The goal of this clinical trial is to learn if the Huandao Conditioning Application works to treat allergic rhinitis in adults. It will also learn about the safety of this application. The main questions it aims to answer are:

Does the Huandao Conditioning Application improve allergic rhinitis symptoms as measured by the Rhinitis Control Assessment Test (RCAT) and nasal airway resistance tests? What medical problems do participants have when using the Huandao Conditioning Application?

Researchers will compare the therapeutic version of the application to a placebo version (a look-alike application that contains no therapeutic effect) to see if the Huandao Conditioning Application works to treat allergic rhinitis.

Participants will:

Use either the therapeutic or placebo version of the application daily for 1 week in Phase 1 Take a 2-week break with no application use Use the opposite version of the application daily for 1 week in Phase 2 Visit the clinic at the beginning and end of each phase for checkups and tests Complete symptom assessment questionnaires before each application use and 1-2 hours after use Be monitored for any adverse reactions throughout the study period

DETAILED DESCRIPTION:
Detailed Description:

Allergic rhinitis (AR) is a chronic respiratory condition affecting 15% of the global population. The study investigates a novel mobile application-based intervention utilizing Traditional Chinese Medicine (TCM) meridian theory.

Study Design:

Randomized, double-blind, placebo-controlled crossover trial Two 1-week treatment periods separated by 2-week washout 1:1 randomization to active/placebo app sequence

Intervention Details:

Therapeutic app: Energy-balancing effects based on TCM meridians Placebo app: Visually identical without therapeutic properties Daily 5-10 minute self-administered sessions Symptom tracking before and 1-2 hours post-application

Assessment Schedule:

Baseline: RCAT, allergen screening, nasal resistance Treatment weeks: Daily symptom monitoring, Day 4 phone follow-up End of phases: RCAT, nasal resistance, adverse events Study completion: Additional allergen screening

Target Population:

95 participants Recruitment via posters at Hualien Tzu Chi Hospital Expected 70 evaluable subjects for analysis

This study aims to evaluate the efficacy and safety of a TCM-based digital therapeutic for AR symptom management.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* RCAT score < 21
* Positive allergen screening (> 0.35 KU/L for house dust, microbial, or pet dander)
* Capable of operating mobile app and completing follow-up

Exclusion Criteria:

* Recent diagnosis, active treatment, or recurrence risk of head/neck cancer
* Current or previous immunotherapy
* Any condition that may compromise participant safety or interfere with trial assessment per investigator judgment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
RCAT scores | Change in RCAT scores [Time Frame: 4 weeks] Baseline (Day 1) End of Phase 1 (Day 8) Start of Phase 2 (Day 22) End of study (Day 29)
  Change in RCAT scores from baseline

SECONDARY OUTCOMES:
Change in nasal airway resistance | Each phase Day 1 and Day 8
  Changes in nasal airway resistance measured by rhinomanometry

IPD SHARING:
Plan to Share IPD: No